CLINICAL TRIAL: NCT02152514
Title: Randomized Controlled Trial Comparing Post-VATS Analgesia Between Patients With an Intrathecal Injection of Morphine and Sufentanil Versus Placebo.
Brief Title: RCT Comparing Analgesia Post-VATS With Epimorph VS Placebo
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to technical details recruitment was unreasonably slow
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Yanick Sansoucy, Anesthesiologist, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Epimorph for VATS
Record Dates: First submitted 2014-05-23; First posted 2014-06-02 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Thoracic Surgery, Video-assisted; Postoperative Pain; Rachianesthesia; Sufentanil; Morphine
MeSH Terms: conditions — Pain, Postoperative | interventions — Sufentanil; Passive Cutaneous Anaphylaxis; Analgesia, Patient-Controlled

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intrathecal Morphine/Sufentanil and PCA (Active Comparator): Patients will receive an intrathecal injection of Morphine 250 mcg and Sufentanil 10 mcg before the induction of anesthesia. They will have a PCA for analgesia rescue in the post-operative period.
  Interventions: Drug: Intrathecal Morphine/Sufentanil; Device: PCA
- PCA alone (Placebo Comparator): Patients will NOT receive an intrathecal injection of Morphine 250 mcg and Sufentanil 10 mcg before the induction of anesthesia. They will only have a PCA for analgesia in the post-operative period.
  Interventions: Device: PCA

INTERVENTIONS:
Drug: Intrathecal Morphine/Sufentanil
  Arms: Intrathecal Morphine/Sufentanil and PCA
Device: PCA
  Other Names: Patient Controlled Analgesia

SUMMARY:
The purpose of the study is to determine if the administration of a mix of Sufentanil and Morphine in intrathecal is a better analgesia regimen than PCA alone in patient post-VATS.

DETAILED DESCRIPTION:
This study will compare the need for analgesia (Hydromorphone PCA) of two groups of patients post-VATS. The placebo group will only have a PCA for post-operative analgesia, witch is the standard care for patient post-VATS. The experimental group will have a intrathecal injection of a mix of morphine and sufentanil before the induction of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* VATS
* ASA 1,2 or 3
* Minimum weight of 50 kg
* Patient able to consent

Exclusion Criteria:

* Patient refusal
* Patient unable to understand PCA
* Contraindication to rachianalgesia
* Zona
* Pregnancy
* Over 30 mg of morphine during the last 24 hours
* Use of Pregabalin, Gabapentin, Doluxetin, Amitriptyline or NSAI in a context of chronic pain
* Severe allergic reaction to morphine, hydromorphone, sufentanil or local anesthetic
* Intubation over 1 hour after surgery (unability to use PCA)
* High risk of conversion to thoracotomy
* Unable to perform rachianalgesia due to technical difficulties

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Hydromorphone consommation | 24hr
  The amount of Hydromorphone needed by the patient in the first 24hr after his VATS.

SECONDARY OUTCOMES:
Pain | Every 4h x 24hr
  A VAS will be used.
Adverse effects of narcotics | Every 4h x 24hr
  Including :
  * Saturation [Saturation (%) and the need for oxygen (l/min) will be assess to evaluate the incidence of desaturation and hypoventilation in both arms]
  * Sedation [Sedation will be evaluate with the Riker Sedation Agitation Scale]
  * Respiratory rate [To evaluate the incidence of hypoventilation (<8/min) and to compare the average between both arms]
Adverse reactions associate with rachianesthesia | 24hr
  Including :
  * Backache
  * Headache
  * Legs strength
Adverse reactions of narcotics | 24hr
  Including :
  * Nausea
  * Pruritis
  * Urinary retention

CONTACTS AND LOCATIONS:
Overall Officials: Yanick Sansoucy, Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Locations (1):
- Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec, Canada